CLINICAL TRIAL: NCT05987878
Title: Single Minimal Conjunctival Incision for Rectus Muscles
Brief Title: Single Minimal Conjunctival Incision for Strabismus
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Jaime Tejedor, Principal Investigator, Universidad Autonoma de Madrid
Other Study IDs: SMCI-22-0213
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Strabismus, Comitant
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: single minimal conjunctival incision — A 5-0 PGA traction suture was used near the corneal limbus corresponding to the operated muscle. A 3-4 mm single conjunctival incision posterior and parallel to the insertion in medial, lateral or superior rectus muscle was used. A hang-back recession of the muscle was done using 6-0 PGA suture. The conjunctiva was closed by an 8-0 PGA single stitch with knot burial

SUMMARY:
The purpose of this investigation is to study the feasibility and inflammatory response of surgery for rectus muscles using a small single bulbar conjunctival incision posterior and parallel to the muscle insertion.

Patients requiring surgery of at least one rectus muscle with several diagnoses, operated under general or topical / sub-Tenon's anesthesia, who had no previous eye muscle surgery, will be recruited. Routinary clinical ophthalmological examination will be carried out. After applying a 5-0 PGA traction suture, a 3-4 mm single conjunctival incision posterior and parallel to the rectus muscle insertion will be done. A hang-back recession with 6-0 PGA suture will be carried out, and the conjunctiva closed by an 8-0 PGA single stitch. The main outcome measure will be duration of swelling and hemorrhage, and secondary outcome measure will be motor outcome at 2 months after surgery.

DETAILED DESCRIPTION:
Purpose/Background: To study the feasibility and inflammatory response of surgery for rectus muscles using a small single bulbar conjunctival incision posterior and parallel to the muscle insertion.

Methods: Patients requiring surgery of at least one rectus muscle with several diagnoses, operated under general or topical / sub-Tenon's anesthesia, who had no previous eye muscle surgery, are included. Routinary clinical ophthalmological examination is carried out. After applying a 5-0 PGA traction suture, a 3-4 mm single conjunctival incision posterior and parallel to the rectus muscle insertion will be done. A hang-back recession with 6-0 PGA suture will be carried out, and the conjunctiva closed by an 8-0 PGA single stitch. The main outcome measure is duration of swelling and hemorrhage, and secondary outcome measure is motor outcome at 2 months after surgery. Results are compared with retrospectively collected data of patients operated using limbal (n= 20) and fornix incision (n= 21) as a point of reference.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring surgery of at least one rectus muscle with several diagnoses, operated under general or topical / sub-Tenon's anesthesia

Exclusion Criteria:

* patients had no previous eye muscle surgery

Ages: 6 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: 25 subjects who required surgery of rectus muscle in comitant strabismus
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Duration of conjunctival swelling/hemorrhage | 2 months
  Evaluate duration of conjunctival swelling/hemorrhage

SECONDARY OUTCOMES:
Motor outcome at 2 months after surgery (by Prism and Alternate Cover Test) | 2 months
  Evaluate motor status at 2 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Tejedor, MD, PhD, Principal Investigator — Universite Abdou Moumouni de Niamey, Niger
Locations (1):
- UAM, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Data shared when solicited to the PI